CLINICAL TRIAL: NCT00007215
Title: A Study of Age-Related Changes in the Human Lens and Cataracts In Vivo Using Dynamic Light Scattering Device (DLS) Combined With Keratoscopy
Brief Title: Dynamic Light Scattering Device (DLS) Study of Age-Related Changes in the Lens and Cataracts
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010051; 01-EI-0051
Record Dates: First submitted 2000-12-15; First posted 2000-12-18 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-02

CONDITIONS: Cataract; Healthy
Keywords: Cataract; Early Lens Changes; Protein Aggregation; Blindness; Vision; Dynamic Laser Scattering (DLS); Age-Related Changes; Test Re-test Reproducibility; Normal Volunteers; Lens; Healthy Volunteer
MeSH Terms: conditions — Cataract; Blindness

SUMMARY:
This study will use a newly developed instrument called dynamic light scattering device (DLS) to examine age-related changes in the human lens and to study the causes and development of cataracts. DLS uses a low intensity laser light (similar to that used in supermarket checkouts) to measures lens cloudiness. It detects changes in the human lens at the earliest stages, when anti-cataract treatment would be most effective in reversing, delaying or preventing cataract formation.

Patients 18 years of age and older with cataracts and normal volunteers between the ages of 18 and 70 years may be eligible for this study. Participants will have a standard eye examination, including a vision check, pressure measurement, lens examination using DLS and examination of the retina. Photographs of the lens or retina, or both, may be taken.

This study does not involve treatment. No anti-cataract medications will be given.

DETAILED DESCRIPTION:
Recently, a device has been created to determine molecular interactions that occur in the nucleus of the lens, called Dynamic Light Scattering Device (DLS). Preliminary studies have shown its potential in the detection of the earliest changes occurring in cataract, at the stage where anticataract treatment would theoretically be most effective in reversing, delaying or preventing cataracts. A new miniaturized version of this device has been developed by NASA using lower energy lasers and offered for further development and testing at the NEI. We recently conducted a pilot study to evaluate the usefulness and reproducibility of this instrument for quantitating lens changes, and found good reproducibility. We also determined that the most useful parameter to use is mean particle size derived from particle size distribution. We therefore propose to conduct a study on changes on the lens due to aging (age related changes), as well as on the three representative types of cataracts (nuclear, cortical and PSC).

ELIGIBILITY:
INCLUSION:

Patients 18 years or older will be admitted to this study.

There will be no gender or sex bias in the recruitment.

Fifteen subjects (30 eyes) who are normal volunteers of either sex, 3 for each decade from 18-70, will be recruited.

These normal volunteers should have clear lenses with LOCS II clinical score for nuclear opalescence of 0.5 or less.

Three patients (18 eyes) for each major type of cataract (nuclear, cortical and PSC), will be recruited also for evaluation with the DLS device.

All 3 types of cataracts will be graded using the LOCS II system and will have a clinical score of at least one.

EXCLUSION:

Patients who have uveitis, glaucoma and who are thought to be at risk for an adverse reaction to pupil dilation, or have a history of allergic reaction to one of the dilating agents that will be used.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 2000-12; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Benedek GB, Chylack LT Jr, Libondi T, Magnante P, Pennett M. Quantitative detection of the molecular changes associated with early cataractogenesis in the living human lens using quasielastic light scattering. Curr Eye Res. 1987 Dec;6(12):1421-32. doi: 10.3109/02713688709044506. PMID 3427992
- [Background] Bursell SE, Baker RS, Weiss JN, Haughton JF, Rand LI. Clinical photon correlation spectroscopy evaluation of human diabetic lenses. Exp Eye Res. 1989 Aug;49(2):241-58. doi: 10.1016/0014-4835(89)90094-8. PMID 2767171
- [Background] Chylack LT Jr, Leske MC, McCarthy D, Khu P, Kashiwagi T, Sperduto R. Lens opacities classification system II (LOCS II). Arch Ophthalmol. 1989 Jul;107(7):991-7. doi: 10.1001/archopht.1989.01070020053028. PMID 2751471